CLINICAL TRIAL: NCT06667089
Title: Comparison of Povidone-Iodine and Chlorhexidine in the Management of Iatrogenic Wounds in Surgical Patients
Brief Title: Povidone-Iodine Versus Chlorhexidine in Surgical Wound Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén¨
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries | interventions — Povidone-Iodine; Chlorhexidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone-Iodine Group (Experimental): The povidone-iodine group will receive applications of 10% povidone-iodine solution or gel directly on the wound area involving a gentle cleaning of the wound followed by the application of povidone-iodine left on for a brief period to maximize its antimicrobial action with treatment applied according to protocol frequency, such as twice daily or as clinically indicated, with close monitoring for any adverse reactions or signs of infection
  Interventions: Other: Povidone-Iodine
- Chlorhexidine Group (Experimental): The chlorhexidine group will receive applications of chlorhexidine solution, typically at a concentration of 0.5% to 2%, also following a gentle cleaning of the wound area before applying chlorhexidine, which will remain on the wound according to protocol guidelines with a similar frequency and monitoring approach to assess for antimicrobial effectiveness, wound healing progress, and potential skin irritation
  Interventions: Other: Chlorhexidine

INTERVENTIONS:
Other: Povidone-Iodine — The povidone-iodine group will receive a 10% povidone-iodine solution or gel applied directly to the wound after gentle cleaning, with the treatment applied according to a set frequency, typically twice daily. This antiseptic will be left on the wound for a brief period to enhance its antimicrobial action.
  Arms: Povidone-Iodine Group
Other: Chlorhexidine — The chlorhexidine group will receive a chlorhexidine solution, usually at a concentration of 0.5% to 2%, applied similarly after cleaning the wound. This solution will remain on the wound according to protocol guidelines, also typically applied twice daily. Both groups will be monitored for adverse reactions, signs of infection, and the overall effectiveness of wound healing throughout the treatment period.
  Arms: Chlorhexidine Group

SUMMARY:
This comparison examines the effectiveness of povidone-iodine and chlorhexidine in managing iatrogenic wounds in surgical patients. Both antiseptics are commonly used to prevent postoperative infections, but they differ in mechanism, efficacy, and safety profiles. Povidone-iodine releases iodine, which acts broadly against bacteria, viruses, and fungi, while chlorhexidine disrupts cell membranes, providing rapid bactericidal action. Studies suggest that chlorhexidine may offer longer-lasting antibacterial effects, but povidone-iodine has a wider antimicrobial range. Optimal choice depends on patient needs, wound type, and potential for adverse reactions, emphasizing the need for tailored antiseptic strategies in wound care.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients undergoing surgical procedures resulting in iatrogenic wounds (surgical wounds of various specialties, such as abdominal, orthopedic, cardiovascular, etc.).
* Availability for follow-up during the postoperative period, ensuring attendance at medical check-ups for the evaluation of healing and prevention of infections.
* Ability to provide informed consent, understanding the objectives, risks and benefits of the study.
* Absence of previous infections at the surgical site, ensuring that the wounds are recent and derived from the current surgical procedure.

Exclusion Criteria:

* Known allergies or hypersensitivity to povidone iodine or chlorhexidine, to avoid risks of serious adverse reactions.
* Immunocompromised patients, such as those with advanced HIV, on immunosuppressant treatment, or with decompensated chronic diseases (poorly controlled diabetes, kidney failure, etc.), due to increased susceptibility to infections and altered healing.
* Patients with active infections or infected wounds prior to surgery, to avoid biasing the results by pre-existing infections.
* Pregnancy or breastfeeding, due to safety considerations and the possible alteration of healing and immunity processes during these stages.
* Use of other antiseptics or topical treatments at the wound site that may interfere with the efficacy of povidone iodine or chlorhexidine.
* Patients with known wound healing disorders (such as autoimmune diseases or hematological disorders), which may affect the results in terms of healing time and quality.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Up to twelve weeks
  The Numerical Rating Scale is a pain assessment tool where patients rate their pain intensity on a scale from 0 to 10, with 0 indicating "no pain" and 10 representing "the worst possible pain." The interpretation of the scores is categorized into levels of pain severity: a score of 0-3 denotes mild pain, 4-6 indicates moderate pain, and 7-10 reflects severe pain. This categorization allows healthcare providers to gauge the patient's pain experience effectively, guiding treatment decisions and evaluating the efficacy of pain management strategies.
EuroQol-5D (EQ-5D) | Up to twelve weeks
  The EuroQol-5D is a standardized instrument for measuring health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The results yield a single index score that typically ranges from -0.594 (worse than death) to 1 (optimal health). Scores are interpreted as follows: 0.0 signifies an average quality of life, 0.5 to 0.8 indicates moderate impairment, and 0.9 to 1.0 reflects high quality of life. These scores are essential for assessing the impact of interventions on patient quality of life.
Patient Satisfaction Questionnaire (PSQ) | Up to twelve weeks
  The Patient Satisfaction Questionnaire assesses patient satisfaction with healthcare services, using a scale from 1 to 5, where 1 represents "very dissatisfied" and 5 indicates "very satisfied." Interpretation of the scores categorizes satisfaction levels: 1-2 denotes low satisfaction, 3 represents average satisfaction, and 4-5 indicates high satisfaction. Higher scores suggest improvements in service quality and patient care, providing valuable feedback for healthcare providers to enhance their practices.
Wound Healing Assessment Tool | Up to twelve weeks
  This tool encompasses various metrics for evaluating wound characteristics, such as size, depth, and signs of infection. Interpretation of the results varies depending on the specific metrics used, but generally, a decrease in wound size and the absence of infection signs signify effective healing. Conversely, the presence of necrosis or an increase in wound size may indicate complications. Higher scores typically correlate with better healing outcomes, guiding clinicians in treatment decisions and monitoring progress.
Adverse Event Reporting Form | Up to twelve weeks
  This form is used to document any adverse reactions or events experienced by patients during treatment. The results are analyzed to calculate the incidence rate of adverse events, with lower rates suggesting that the treatment is safe and well-tolerated. Conversely, a higher frequency of adverse events may indicate safety concerns, prompting further investigation and potential modifications in treatment protocols. These findings are critical for evaluating the safety profile of interventions and informing clinical practice.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Up to twelve weeks
  Assesses symptoms of anxiety and depression using 14 items (7 for each subscale), each scored from 0 to 3. Scores range from 0 to 21 for anxiety and for depression, where 0-7 is normal, 8-10 indicates possible symptoms, and 11 or higher suggests a clinical disorder.
Pittsburgh Sleep Quality Index (PSQI) | Up to twelve weeks
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result. Higher scores indicate poorer sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- María Juana Millán Reyes, Jaén, Spain